CLINICAL TRIAL: NCT06679244
Title: Application of Hao's Esophagogastrostomy by Fissure Technique: a Prospective, Multicenter Randomized Controlled Study
Brief Title: Application of a New Surgical Technique in Proximal Gastrectomy: a Prospective, Multicenter Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Cancer Hospital, China (Other)
Responsible Party: Principal Investigator, Hao Hankun, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1173
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer Patients Undergoing Minimally Invasive Gastrectomy
Keywords: proximal gastrectomy; totally laparoscopic gastrectomy; fissure technique

STUDY DESIGN:
Intervention Model Description: Based on the different anastomotic methods used in proximal gastrectomy, patients are divided into a HEFT group (experimental group) and a double-tract reconstruction group (control group).
  HEFT group:Patients included in this group will receive totally laparoscopic proximal gastrectomy with Hao's esophagogastrostomy by fissure technique(HEFT)，which is an innovative surgery that investigators first began to apply in patients with proximal gastric cancer.
  double-tract reconstruction group:Patients included in this group will receive totally laparoscopic proximal gastrectomy with double-tract reconstruction group，which is a widely used and proven safe and effective surgical approach in proximal gastrectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Performing Hao's esophagogastrostomy by fissure technique (Experimental)
  Interventions: Procedure: Totally laparoscopic proximal gastrectomy with Hao's esophagogastrostomy by fissure technique
- Performing double-tract reconstruction (Active Comparator)
  Interventions: Procedure: Totally laparoscopic proximal gastrectomy with double-tract reconstruction

INTERVENTIONS:
Procedure: Totally laparoscopic proximal gastrectomy with Hao's esophagogastrostomy by fissure technique — This is an innovative surgical method applied in proximal gastrectomy. By adding anti reflux structures such as "false gastric fundus" and "false cardia" on the basis of esophageal residual gastric anastomosis, the goal of anti reflux is achieved, while maintaining normal physiological channels and fully utilizing residual gastric function, reducing the difficulty of proximal gastrectomy surgery
  Arms: Performing Hao's esophagogastrostomy by fissure technique
Procedure: Totally laparoscopic proximal gastrectomy with double-tract reconstruction — This is a traditional surgical method that has been widely used in proximal gastrectomy. After disconnecting the proximal stomach, performing Roux-en-Y anastomosis of the esophagus and jejunum firstly, followed by lateral anastomosis of the residual stomach and jejunum. Previous studies have confirmed its safety and effectiveness, but there are also issues of gastric channel disuse and high missed detection rate of residual stomach.
  Arms: Performing double-tract reconstruction

SUMMARY:
This is a prospective study using a multicenter, randomized, controlled, open label, and efficacy validated approach.At present, there is no universally recognized optimal method for gastrointestinal reconstruction after proximal gastrectomy in the surgical treatment of gastric cancer.Author's team has proposed an innovative method named Hao's Esophagogastrostomay by Fisture Technique (HEFT).By adding anti reflux structures such as "false gastric fundus" and "false cardia" to the anastomosis of the residual stomach of the esophagus, not only can the purpose of anti reflux be achieved, but also the normal physiological channel can be maintained, it can fully utilize residual stomach function and reduce the difficulty of surgery.Through retrospective research, our single center has confirmed that HEFT is safe and feasible.On this basis, this study will compare the nutritional status, short- and medium- to long-term safety after laparoscopic HEFT and double-tract reconstruction , in order to evaluate and discover more reasonable digestive tract reconstruction methods after proximal gastrectomy, and to promote the development and popularization of minimally treatment technology for gastric cancer.

This study was jointly conducted by Shanghai-level hospitals (Huashan Hospital ,Shanghai Cancer Center, and Ruijin Hospital), with Huashan Hospital as the leading unit. This study will recruit 52 patients, with 26 patients in the experimental group and 26 patients in the control group. Using a central dynamic randomization method based on minimization, patients are assigned to groups in a 1:1 ratio. Based on the different anastomotic methods used in proximal gastrectomy, patients are divided into a HEFT group (experimental group) and a double-tract reconstruction group (control group).Plan to collect cases for 2 years, and follow up for another year after the last case is enrolled.

The primary endpoint of the study was the body weight loss (BWL) rate at 1 year after surgery. Secondary endpoints: Effect evaluation indicators: hemoglobin level at 1 year after surgery; Serum albumin level at 1 year after surgery; The incidence of anastomotic stenosis 1 year after surgery; Incidence of reflux esophagitis at 1 year after surgery. Evaluation of short-term surgical safety (duration: 7 days): operation time, intraoperative bleeding, anastomotic leakage, pancreatic leakage, and incidence of abdominal infection; Evaluation of medium- and long-term safety after surgery (duration: 36 months): overall survival rate at 3 years after surgery; disease-free survival rate at 3 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ 80 years old;
2. The primary tumor lesion is located in the upper part of the stomach or the esophagogastric junction (Siewert II or III), and it is expected that R0 surgical results can be obtained by performing proximal gastrectomy and D2 dissection；
3. The primary lesion was diagnosed as adenocarcinoma through endoscopic biopsy and histopathological examination;
4. If it is upper gastric adenocarcinoma, the clinical TNM staging based on imaging needs to be cT1N0M0. If it is ductal gastric junction adenocarcinoma, it needs to be cT1-3N0-1M0, and clinical imaging judgment shows no distant gastric lymph node metastasis；
5. Expected survival exceeds 6 months;
6. No history of upper abdominal surgery (excluding laparoscopic cholecystectomy);
7. No chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc. were performed before surgery;
8. Preoperative ECOG (Eastern Cooperative Oncology Group) physical status score 0/1;
9. Preoperative ASA (American Society of Anesthesiologists) grading I-III ;
10. Good function of important organs;
11. Sign the patient's informed consent form

Exclusion Criteria:

1. Preoperative imaging examination suggests the fusion of enlarged lymph nodes (maximum diameter ≥ 3cm) in the area;
2. Pregnant and lactating women;
3. Suffering from other malignant tumors within 5 years;
4. Preoperative body temperature ≥ 38 ℃ or complicated with infectious diseases requiring systematic treatment;
5. Serious mental illness;
6. Severe respiratory diseases, FEV1<50% of the expected value;
7. Severe liver and kidney dysfunction;
8. History of unstable angina or heart attack within 6 months;
9. History of cerebral infarction or cerebral hemorrhage within 6 months, excluding old intracavitary infarction;
10. Apply systemic corticosteroid therapy within one month;
11. Patients with complications of gastric cancer (bleeding, perforation, obstruction) requiring emergency surgery;
12. The patient has participated or is currently participating in other clinical studies (within 6 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
body weight loss（BWL） | From enrollment to 1 year after surgery
  Measure the weight before surgery and 1 year after surgery, BWL=(preoperative weight -1 year after surgery weight)/preoperative weight (unit:%)

SECONDARY OUTCOMES:
Hemoglobin 1 year after surgery | 1 year after surgery
  Hemoglobin (unit: g/L) 1 year after surgery will be used to evaluate operation effect.
Serum albumin 1 year after surgery | 1 year after surgery
  Serum albumin (unit: g/L) 1 year after surgery will be used to evaluate operation effect.
Incidence of anastomotic stenosis 1 year after surgery | 1 year after surgery
  Incidence of anastomotic stenosis(%) 1 year after surgery will be used to evaluate operation effect.
Incidence of reflux esophagitis 1 year after surgery | 1 year after surgery
  Incidence of reflux esophagitis 1 year after surgery will be used to evaluate operation effect.
Duration of surgery | intraoperative
  Time spent on the whole operation（minutes）will be used to evaluate short-term safety of the surgery
Intraoperative blood loss | Intraoperative
  Intraoperative blood loss(ml) will be used to evalute short-term safety of the surgery.
Incidence of anastomotic leakage 7 days after surgery | 7 days after surgery
  Incidence of anastomotic leakage(%) 7 days after surgery will be used to evaluate short-term safety of the surgery
Incidence of pancreatic leakage 7 days after surgery | 7 days after surgery
  Incidence of pancreatic leakage 7 days after surgery will be used to evaluate short-term safety of the surgery.
Incidence of abdominal infection 7 days after surgery | 7 days after surgery
  Incidence of abdominal infection 7 days after surgery will be used to evaluate short-term safety of the surgery.
Overall survival (OS) 3 years after surgery | 3 years after surgery
  Overall survival (OS, %) 3 years after surgery will be used to evaluate medium- and long-term postoperative safety
Disease free survival (DFS) 3 years after surgery | 3 years after surgery
  Disease free survival (DFS, %) 3 years after surgery will be used to evaluate medium- and long-term postoperative safety,

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Department of General Surgery, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - Second Department of Gastric Surgery, Fudan University Shanghai Cancer Center,, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sakuramoto S, Yamashita K, Kikuchi S, Futawatari N, Katada N, Moriya H, Hirai K, Watanabe M. Clinical experience of laparoscopy-assisted proximal gastrectomy with Toupet-like partial fundoplication in early gastric cancer for preventing reflux esophagitis. J Am Coll Surg. 2009 Sep;209(3):344-51. doi: 10.1016/j.jamcollsurg.2009.04.011. Epub 2009 Jun 18. PMID 19717038
- [Background] Aizawa M, Yabusaki H, Nakada K, Matsuki A, Bamba T, Nakagawa S. A Retrospective Review of a Single-Center Experience with Posterolateral Fundoplication During Esophagogastrostomy After Proximal Gastrectomy. J Gastrointest Surg. 2021 Dec;25(12):3230-3233. doi: 10.1007/s11605-021-05052-8. Epub 2021 Jul 8. No abstract available. PMID 34240326
- [Background] Shoji Y, Nunobe S, Ida S, Kumagai K, Ohashi M, Sano T, Hiki N. Surgical outcomes and risk assessment for anastomotic complications after laparoscopic proximal gastrectomy with double-flap technique for upper-third gastric cancer. Gastric Cancer. 2019 Sep;22(5):1036-1043. doi: 10.1007/s10120-019-00940-0. Epub 2019 Mar 6. PMID 30838469
- [Background] Kuroda S, Choda Y, Otsuka S, Ueyama S, Tanaka N, Muraoka A, Hato S, Kimura T, Tanakaya K, Kikuchi S, Tanabe S, Noma K, Nishizaki M, Kagawa S, Shirakawa Y, Kamikawa Y, Fujiwara T. Multicenter retrospective study to evaluate the efficacy and safety of the double-flap technique as antireflux esophagogastrostomy after proximal gastrectomy (rD-FLAP Study). Ann Gastroenterol Surg. 2018 Oct 11;3(1):96-103. doi: 10.1002/ags3.12216. eCollection 2019 Jan. PMID 30697614
- [Background] Aihara R, Mochiki E, Ohno T, Yanai M, Toyomasu Y, Ogata K, Ando H, Asao T, Kuwano H. Laparoscopy-assisted proximal gastrectomy with gastric tube reconstruction for early gastric cancer. Surg Endosc. 2010 Sep;24(9):2343-8. doi: 10.1007/s00464-010-0947-8. Epub 2010 Apr 8. PMID 20376493
- [Background] Tanaka K, Ebihara Y, Kurashima Y, Nakanishi Y, Asano T, Noji T, Murakami S, Nakamura T, Tsuchikawa T, Okamura K, Shichinohe T, Hirano S. Laparoscopic proximal gastrectomy with oblique jejunogastrostomy. Langenbecks Arch Surg. 2017 Sep;402(6):995-1002. doi: 10.1007/s00423-017-1587-4. Epub 2017 May 10. PMID 28493146
- [Background] Aikou T, Natsugoe S, Shimazu H, Nishi M. Antrum preserving double tract method for reconstruction following proximal gastrectomy. Jpn J Surg. 1988 Jan;18(1):114-5. doi: 10.1007/BF02470857. PMID 3386066
- [Background] Zang L. [Reconstruction following laparoscopic gastrectomy for gastric cancer]. Zhonghua Wei Chang Wai Ke Za Zhi. 2012 Aug;15(8):787-9. Chinese. PMID 23072016
- [Background] Fujiya K, Kawamura T, Omae K, Makuuchi R, Irino T, Tokunaga M, Tanizawa Y, Bando E, Terashima M. Impact of Malnutrition After Gastrectomy for Gastric Cancer on Long-Term Survival. Ann Surg Oncol. 2018 Apr;25(4):974-983. doi: 10.1245/s10434-018-6342-8. Epub 2018 Jan 31. PMID 29388124
- [Background] Yamasaki M, Takiguchi S, Omori T, Hirao M, Imamura H, Fujitani K, Tamura S, Akamaru Y, Kishi K, Fujita J, Hirao T, Demura K, Matsuyama J, Takeno A, Ebisui C, Takachi K, Takayama O, Fukunaga H, Okada K, Adachi S, Fukuda S, Matsuura N, Saito T, Takahashi T, Kurokawa Y, Yano M, Eguchi H, Doki Y. Multicenter prospective trial of total gastrectomy versus proximal gastrectomy for upper third cT1 gastric cancer. Gastric Cancer. 2021 Mar;24(2):535-543. doi: 10.1007/s10120-020-01129-6. Epub 2020 Oct 29. PMID 33118118
- [Background] Japanese Gastric Cancer Association. Japanese Gastric Cancer Treatment Guidelines 2021 (6th edition). Gastric Cancer. 2023 Jan;26(1):1-25. doi: 10.1007/s10120-022-01331-8. Epub 2022 Nov 7. PMID 36342574
- [Background] GBD 2017 Stomach Cancer Collaborators. The global, regional, and national burden of stomach cancer in 195 countries, 1990-2017: a systematic analysis for the Global Burden of Disease study 2017. Lancet Gastroenterol Hepatol. 2020 Jan;5(1):42-54. doi: 10.1016/S2468-1253(19)30328-0. Epub 2019 Oct 21. PMID 31648970
- [Derived] Cui WL, Wang ZQ, Shi XL, Ma MY, Wang J, Wang ZH, Wang YP, Hong J, Hao HK. Application of Hao's Esophagogastrostomy by Fissure Technique (HEFT) in proximal gastrectomy: protocol for a prospective, multicentre, randomised controlled study. BMJ Open. 2025 Aug 12;15(8):e104365. doi: 10.1136/bmjopen-2025-104365. PMID 40803728